CLINICAL TRIAL: NCT03552965
Title: Prospective Randomized Pilot Clinical Trial of Margin-Based Vs. Robust Photon Radiotherapy Planning in Intensity-Modulated Radiation Therapy of Squamous-Cell Carcinoma of the Head and Neck
Brief Title: Margin-Based Vs. Robust Photon Radiotherapy Planning in IMRT of HN-SQCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 217585
Record Dates: First submitted 2018-05-07; First posted 2018-06-12 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: xerostomia; Robust photon radiotherapy; Margin based radiotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Margin-Based Radiotherapy Planning (Active Comparator): This arm will receive Intensity-Modulated Radiation Therapy (IMRT) that was calculated by introducing a margin to the target area.
  Interventions: Other: Margin-Based Radiotherapy planning
- Robust Radiotherapy Planning (Active Comparator): This arm will receive Intensity-Modulated Radiation Therapy (IMRT) that was calculated to minimize the dose of radiation to normal tissue.
  Interventions: Other: Robust Radiotherapy planning

INTERVENTIONS:
Other: Robust Radiotherapy planning — Investigator will plan Intensity-Modulated Radiation Therapy (IMRT) using calculations that minimize the dose of radiation to normal tissue
  Arms: Robust Radiotherapy Planning
Other: Margin-Based Radiotherapy planning — Investigator will plan Intensity-Modulated Radiation Therapy (IMRT) using calculations that introduce a margin to the target area
  Arms: Margin-Based Radiotherapy Planning

SUMMARY:
This is a research study to evaluate the quality of life and amount of dry mouth experienced as a result of radiotherapy in subjects who have squamous cell carcinoma of the head and neck (HN-SQCC). This study will compare the side effects experienced based on the method to plan radiotherapy, Margin Based or Robust.

DETAILED DESCRIPTION:
This is a prospective randomized pilot clinical trial, stratified by primary tumor site, to evaluate the degree of xerostomia and quality of life (QOL) in subjects with HN-SQCC treated with radiation therapy under margin-based and robust radiotherapy treatment plans. Margin-based plans will use both biological (biological optimization) and physical objectives whereas robust planning will use physical objectives for sparing of the parotid glands. Intensity-modulated radiation therapy (IMRT) and standard chemotherapy will be used. QOL (quality of life) will be measured using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 questionnaire and EORTC QLQ-H&N35 (head and neck) module before radiotherapy (baseline) and then 3, 6, 9 and 12 months after radiotherapy. Xerostomia will be measured in study subjects using two patient-reported scoring systems completed by each subject before radiotherapy and then 3, 6, 9, and 12 months after radiotherapy: Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA) LENT/SOMA grading system and the University of Michigan's Xerostomia Questionnaire (XQ). The data collected by this randomized pilot clinical trial will be used to inform the design of, and decision-making for, future larger studies that seek to compare different methods of radiotherapy planning in the treatment of HN-SQCC.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Squamous-Cell Carcinoma of the Head and Neck (HN-SQCC)
* Older than 21 years of age
* Subject is eligible for routine chemo-radiotherapy for treatment of HN-SQCC
* Informed consent is obtained
* Karnofsky performance of at least 70 points

Exclusion Criteria:

* Women with a positive urine pregnancy test are excluded from this study; women of childbearing potential must agree to refrain from breast feeding and practice adequate contraception
* Unable to comply with study procedures
* Use of saliva stimulating prescription drugs such as Evoxac or Salagen
* Unable to receive standard chemotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2024-03-09 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mausam Patel, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Started | 10 | 13
Completed | 5 | 8
Not Completed | 5 | 5
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Continuation not in patient best interest | 1 | 0
Not completed — Patient opted to be treated elsewhere | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9615 (9.37823) | 62.8215 (11.87871) | 62.8824 (10.62783)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 12 | 20
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23
Late Effects Normal Tissue Task Force-Subjective, Objective, Management, Analytic scale (LENT-SOMA) [Mean (Standard Deviation); unit: units on a scale] — Self reported dry mouth using Late Effects Normal Tissue Task Force -Subjective, Objective, Management, Analytic (LENT/SOMA) scale. LENT/SOMA measures xerostomia in 4 stages. This ranges from Stage 1 "occasional dryness" through Stage 4 "complete dryness, debilitating". Lower stage values indicate a more favorable outcome than higher stage values.
  units on a scale | 1.14 (0.378) | 1.17 (0.577) | 1.16 (0.501)
University of Michigan's Xerostomia Questionnaire (XQ) [Mean (Standard Deviation); unit: score on a scale] | 15.5 (23.76242) | 14.1346 (17.87095) | 14.7283 (20.14139)

OUTCOME MEASURES:

1. Primary Outcome: Grade of Xerostomia
Description: Self reported dry mouth using Late Effects Normal Tissue Task Force -Subjective, Objective, Management, Analytic (LENT/SOMA) scale. LENT/SOMA measures xerostomia in 4 stages. This ranges from Stage 1 "occasional dryness" through Stage 4 "complete dryness, debilitating". Lower stage values indicate a more favorable outcome than higher stage values.
Time Frame: Baseline
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 7 | 12
units on a scale | 1.14 (0.378) | 1.17 (0.577)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=1.14, SD=0.378, Range=1, 25th percentile=1, Median=1, 75th percentile=1, n=7 Robust: Mean=1.17, SD=0.577, Range=2, 25th percentile=1, Median=1, 75th percentile=1, n=12

2. Primary Outcome: Grade of Xerostomia
Description: as for outcome 1
Time Frame: Month 3 (i.e., 3 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 6 | 11
units on a scale | 2.00 (0.894) | 2.91 (1.136)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=2, SD=0.894, Range=2, 25th percentile=1, Median=2, 75th percentile=3, n=6 Robust: Mean=2.91, SD=1.136, Range=3, 25th percentile=2, Median=3, 75th percentile=4, n=11

3. Primary Outcome: Grade of Xerostomia
Description: as for outcome 1
Time Frame: Month 6 (i.e., 6 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 4 | 9
units on a scale | 2.5 (0.577) | 2.33 (1.225)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=2.5, SD=0.577, Range=1, 25th percentile=2, Median=2.5, 75th percentile=3, n=4 Robust: Mean=2.33, SD=1.225, Range=3, 25th percentile=1, Median=2, 75th percentile=3.5, n=9

4. Primary Outcome: Grade of Xerostomia
Description: as for outcome 1
Time Frame: Month 9 (i.e., 9 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 6 | 9
units on a scale | 1.83 (0.753) | 2.33 (1.000)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=1.83, SD=0.753, Range=2, 25th percentile=1, Median=2, 75th percentile=2.25, n=6 Robust: Mean=2.33, SD=1, Range=3, 25th percentile=1.5, Median=2, 75th percentile=3, n=9

5. Primary Outcome: Grade of Xerostomia
Description: as for outcome 1
Time Frame: Month 12 (i.e., 12 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 5 | 8
units on a scale | 2.00 (0.707) | 2.38 (1.188)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=2, SD=0.707, Range=2, 25th percentile=1.5, Median=2, 75th percentile=2.5, n=5 Robust: Mean=2.38, SD=1.188, Range=3, 25th percentile=1.25, Median=2, 75th percentile=3.75, n=8

6. Primary Outcome: Prevalence of Xerostomia
Description: Self reported dry mouth using University of Michigan's Xerostomia Questionnaire (XQ). This questionnaire has 8 questions that measure the degree to which xerostomia is affecting quality of life. Patients rate each item on a scale from 0 to 10. Higher score denotes worse xerostomia. To analyze the XQ, scores on its 8 items will be summed for each subject at each time point to produce an overall XQ score whose values theoretically can range from 0 to 80; it will be treated as a continuous variable. Lower values indicate a more favorable outcome than higher values.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 10 | 13
score on a scale | 15.5 (23.76242) | 14.1346 (17.87095)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=15.5, SD=23.76242, Range=75, 25th percentile=0, Median=5, 75th percentile=21.25, n=10 Robust: Mean=14.1346, SD=17.87095, Range=52.5, 25th percentile=0, Median=6.25, 75th percentile=27.5, n=13

7. Primary Outcome: Prevalence of Xerostomia
Description: as for outcome 6
Time Frame: Month 3 (i.e., 3 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 6 | 11
score on a scale | 45.625 (30.68744) | 64.3182 (15.0142)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=45.625, SD=30.68744, Range=71.25, 25th percentile=11.25, Median=58.125, 75th percentile=71.25, n=6 Robust: Mean=64.3182, SD=15.0142, Range=48.75, 25th percentile=66.25, Median=70, 75th percentile=71.25, n=11

8. Primary Outcome: Prevalence of Xerostomia
Description: as for outcome 6
Time Frame: Month 6 (i.e., 6 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 5 | 9
score on a scale | 60.0000 (23.68412) | 54.8611 (29.91815)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=60, SD=23.68412, Range=60, 25th percentile=38.125, Median=68.75, 75th percentile=77.5, n=5 Robust: Mean=54.8611, SD=29.91815, Range=80, 25th percentile=24.375, Median=66.25, 75th percentile=80, n=9

9. Primary Outcome: Prevalence of Xerostomia
Description: as for outcome 6
Time Frame: Month 9 (i.e., 9 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 6 | 9
score on a scale | 31.6667 (31.38139) | 54.0278 (24.57274)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=31.67, SD=31.38139, Range=85, 25th percentile=5.625, Median=25, 75th percentile=56.875, n=6 Robust: Mean=54.0278, SD=24.57274, Range=67.5, 25th percentile=33.75, Median=62.5, 75th percentile=72.5, n=9

10. Primary Outcome: Prevalence of Xerostomia
Description: as for outcome 6
Time Frame: Month 12 (i.e., 12 months (+/- 30 days) after baseline visit)
Population: There were missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
Number analyzed (Participants) | 5 | 8
score on a scale | 50.75 (30.29284) | 38.4375 (26.69897)
Statistical Analysis 1: Comparison: Margin-Based Radiotherapy Planning vs Robust Radiotherapy Planning; Test type: Other; Descriptive statistics were used to evaluate the prevalence and grade of xerostomia over time. Margin-based: Mean=50.75, SD=30.29284, Range=72.5, 25th percentile=21.875, Median=48.75, 75th percentile=80.625, n=5 Robust: Mean=38.4375, SD=26.69897, Range=66.25, 25th percentile=15, Median=29.375, 75th percentile=68.75, n=8

ADVERSE EVENTS:
Time Frame: Baseline to Month 12 (i.e., 12 months (+/- 30 days) after baseline visit)
Arm/Group | Margin-Based Radiotherapy Planning | Robust Radiotherapy Planning
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/10 | 5/13
Other Adverse Events (participants affected / at risk) | 3/10 | 6/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Margin-Based Radiotherapy Planning (N=10) | Robust Radiotherapy Planning (N=13)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 4 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 1 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (2) | 1 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Margin-Based Radiotherapy Planning (N=10) | Robust Radiotherapy Planning (N=13)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1) | 5 (7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (8) | 5 (8)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 2 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 5 (11)
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (9)
Dysphagia (Gastrointestinal disorders) | 2 (5) | 4 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 6 (8)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3) | 3 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (13) | 3 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (7) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 4 (10)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Investigations - Other, specify (Investigations) | 2 (11) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (6) | 6 (18)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (4)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (9) | 4 (5)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 2 (3)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (6)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5)
Weight loss (Investigations) | 2 (2) | 2 (4)
White blood cell decreased (Investigations) | 1 (1) | 5 (17)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Neck edema (General disorders) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 5 (6)
Scleral disorder (Eye disorders) | 0 (0) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT03552965/Prot_SAP_000.pdf